CLINICAL TRIAL: NCT07401186
Title: Stimulation Evoked Primary Afferent Depolarization to Modulate Sensory Transmission to Spinal Motoneurons and the Sensory Cortex
Brief Title: Stimulation-Based Modulation of Spinal and Cortical Sensory Pathways
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peter C. Gerszten, MD (Other)
Responsible Party: Sponsor-Investigator, Peter C. Gerszten, MD, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY25040076
Record Dates: First submitted 2026-01-29; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Stroke; Able Bodied
Keywords: Central Nervous System Disease; Cerebrovascular Disorder; Brain Injury; Brain Disease; Movement Disorder; Nervous System; Stroke; Spinal Cord Disease; Nervous System Disease; Sensorimotor Disorder
MeSH Terms: conditions — Stroke; Central Nervous System Diseases; Cerebrovascular Disorders; Brain Injuries; Brain Diseases; Movement Disorders; Neurologic Manifestations; Spinal Cord Diseases; Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: This is a prospective, controlled, open-label, experimental study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Dorsal Spinal Nerve Root Stimulation (Experimental): Individuals undergoing cervical spinal surgery will receive direct electrical stimulation to the cervical dorsal spinal nerve roots.
  Interventions: Device: Bipolar Neural Stimulation Electrode

INTERVENTIONS:
Device: Bipolar Neural Stimulation Electrode — All individuals enrolled in this study will receive electrical stimulation to the dorsal cervical spinal nerves using the FDA-cleared bipolar stimulating electrode routinely used as standard-of-care to monitor neural function, during which muscle activities will be recorded through intramuscular electromyography (EMGs), and sensory evoked cortical local field potentials (SSEPs) will be acquired simultaneously to characterize properties of the spinal sensory pathways.

SUMMARY:
The goal of this study is to assess cervical (neck) reflexes by intra-operatively stimulating the neck nerve roots to evoke motor responses through their connections to spinal motoneurons. This data is critical to reveal changes to the spinal sensory modulating circuitry in neurological disorders like stroke.

DETAILED DESCRIPTION:
Spinal afferents continuously convey sensory information on limb movements to the central nervous system which not only gives us conscious experience of movement, but also plays a major role in shaping motor output through monosynaptic afferent-motoneuronal connections. Stroke induces changes in the spinal circuitry modulating this sensory input, leading to sensorimotor deficits.

Specifically, we will 1) activate the dorsal root fibers with single and double electrical stimulation pulses at various frequencies using FDA-cleared devices, 2) quantify the stimulation evoked motor potentials in arm and hand muscles recorded with intramuscular EMGs, 3) quantify stimulation evoked sensory potentials in the cortex with intra-op EEGs.

ELIGIBILITY:
Inclusion Criteria:

* All Subjects: Ages between 21 and 75 years. The minimum age is selected to age match control subjects with stroke subjects. In addition, participants outside this age range may be at an increased medical risk.
* Control subjects: Patients undergoing elective posterior cervical spinal surgery that includes a decompressive laminectomy, and who will have electrophysiological monitoring performed as part of the standard of care for their procedure.
* Stroke subjects: Participants must have a suffered a single, ischemic or hemorrhagic stroke more than 6 months prior to the time of enrollment with hemiparesis as a result, is undergoing a cervical epidural lead implant or undergoing elective posterior cervical spinal surgery that includes a decompressive laminectomy with electrophysiological monitoring performed as part of the standard of care.

Exclusion Criteria:

* Patients will be excluded from the study if they have any known neurological diseases other than stroke, such as amyotrophic lateral sclerosis, spinal muscular atrophy, spinal cord injury, autoimmune neuropathy, or sensory nerve disorders, that may affect the integrity of cervical sensory afferents.
* Only patients that are eligible for surgery will be enrolled. Therefore this automatically include as exclusion criteria: pregnancy and other clinical conditions eligible for surgery.
* Participants must not be on anti-spasticity or anti-epileptic medications.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Spinal Circuit Excitability | 1 day
  The investigators will record intramuscular electromyogram (EMG) of the hand and arm muscles evoked by dorsal nerve root stimulation at various frequencies to quantify spinal circuit excitability through the H-reflex. A mean difference of 10% from the baseline (first pulse per frequency) muscle activation will be considered a meaningful change in excitability.

SECONDARY OUTCOMES:
Sensory Transmission to the Brain | 1 day
  The investigators will use electroencephalograph (EEG) to record sensory stimulation evoked potentials (SSEP) from the brain during dorsal root stimulation at various frequencies to quantify sensory transmission efficiency. A mean difference of 10% from the baseline (first pulse per frequency) SSEP will be considered a meaningful change.

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Gerszten, MD, Principal Investigator — University of Pittsburgh, Neurological Surgery
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification, may be shared with other researchers for the purpose of data analysis and collaboration.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available at the end of the trial upon publication of the first manuscript. Estimation is 5 years from enrollment of the first participant.
Access Criteria: Data must be directly requested from the PI and will be shared upon completion of the necessary data-sharing agreement to protect confidential patient information.